CLINICAL TRIAL: NCT04078295
Title: An Open-Label Phase 1b/2 Study of E7389 Liposomal Formulation Plus Nivolumab in Subjects With Solid Tumor
Brief Title: A Study of E7389 Liposomal Formulation (E7389-LF) Plus Nivolumab in Participants With Solid Tumor
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E7389-J081-120
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Solid Neoplasms
Keywords: E7389 liposomal formulation; Nivolumab; Neoplasms; Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Phase 1b, Cohort 1: E7389-LF Dose 1 + Nivolumab Dose 1 (Experimental): Participants will receive E7389-LF (intravenous) Dose 1 and nivolumab (intravenous) Dose 1 on specified days.
  Interventions: Drug: E7389-LF; Drug: Nivolumab
- Phase 1b, Cohort 2: E7389-LF Dose 2 + Nivolumab Dose 1 (Experimental): Participants will receive E7389-LF (intravenous) Dose 2 and nivolumab (intravenous) Dose 1 on specified days.
  Interventions: Drug: E7389-LF; Drug: Nivolumab
- Phase 1b, Cohort 3: E7389-LF Dose 3 + Nivolumab Dose 2 (Experimental): Participants will receive E7389-LF (intravenous) Dose 3 and nivolumab (intravenous) Dose 2 on specified days.
  Interventions: Drug: E7389-LF; Drug: Nivolumab
- Phase 1b, Cohort 4: E7389-LF Dose 4 + Nivolumab Dose 2 (Experimental): Participants will receive E7389-LF (intravenous) Dose 4 and nivolumab (intravenous) Dose 2 on specified days.
  Interventions: Drug: E7389-LF; Drug: Nivolumab
- Phase 2, Cohort-1: E7389-LF + Nivolumab (Experimental): Participants with gastric cancer will receive RP2D of E7389-LF (intravenous) and nivolumab (intravenous) determined in Phase 1b part.
  Interventions: Drug: E7389-LF; Drug: Nivolumab
- Phase 2, Cohort-2: E7389-LF + Nivolumab (Experimental): Participants with esophageal cancer will receive RP2D of E7389-LF (intravenous) and nivolumab (intravenous) determined in Phase 1b part.
  Interventions: Drug: E7389-LF; Drug: Nivolumab
- Phase 2, Cohort-3: E7389-LF + Nivolumab (Experimental): Participants with small lung cancer will receive RP2D of E7389-LF (intravenous) and nivolumab (intravenous) determined in Phase 1b part.
  Interventions: Drug: E7389-LF; Drug: Nivolumab

INTERVENTIONS:
Drug: E7389-LF — E7389-LF Intravenous infusion.
Drug: Nivolumab — Nivolumab Intravenous infusion.
  Other Names: ONO-4538

SUMMARY:
The primary purpose of the study is to evaluate safety and tolerability of E7389 liposomal formulation (E7389-LF) in combination with nivolumab and to determine the recommended Phase 2 dose (RP2D) in Phase 1b part and to evaluate objective response rate (ORR) of E7389-LF and nivolumab using RP2D in each tumor type in Phase 2 part.

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1b part only: Participants with advanced, nonresectable, or recurrent solid tumor for which no alternative standard therapy or no effective therapy exists (participants who will be the candidate of treatment by nivolumab monotherapy as standard therapy is acceptable)
2. Phase 2 part only: Participants with a confirmed diagnosis of nonresectable gastric cancer (GC), esophageal cancer (EGC) or small cell lung cancer (SCLC) who showed disease progression based on investigator's assessment during or after first line chemotherapy (second-line chemotherapy for GC) and did not receive any other systemic chemotherapy to advanced/recurrent disease
3. Participants who meet the following criteria for biopsy; Phase 1b part: Participants who have accessible tumors for biopsy and agree to tumor biopsy for pre- and post-treatment of study drug (If a pre-treatment biopsy cannot be obtained due to safety issue, then an archival tumor tissue sample may be submitted.) Phase 2 part: Participants who have accessible tumors for biopsy and agree with tumor biopsy for pre and post treatment of study drug (As an alternative to pre-treatment biopsy, tumor tissue sample taken from recurrent or advanced disease may be submitted). However, if the sponsor and the investigator discuss and agree in advance, and the participants agree to submission of archival tumor tissue, then these participants are eligible regardless of accessible tumors, and consent to biopsy is not necessary
4. Life expectancy of greater than or equal to (>=) 12 weeks
5. Eastern Cooperative Oncology Group-Performance Status (ECOG-PS) 0-1
6. Phase 2 part only: At least one measurable lesion based on RECIST 1.1 (Lesions that have had radiotherapy or loco-regional therapies must show evidence of progressive disease to be deemed a measurable lesion)

Exclusion Criteria:

1. Diagnosed with meningeal carcinomatosis
2. Participants with brain or subdural metastases or invasion are not eligible
3. Active, known, or suspected autoimmune disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of Participants with Dose Limiting Toxicities (DLTs) | Baseline up to Cycle 1 (Cycle length is equal to [=] up to 28 days)
  DLTs are defined as study drug related adverse events (AEs). Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE 5.0).
Phase 2: ORR | Baseline up to End of Treatment (Up to approximately 79 months)
  ORR is defined as the percentage of participants who have best overall response of complete response (CR) or partial response (PR). The ORR will be assessed by investigator based on response evaluation criteria in solid tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Phase 1b and Phase 2: Number of Participants With AEs and Serious Adverse Events (SAEs) | Up to 30 days after the last dose of study drug or before initiating post anti-cancer treatment, whichever shorter (up to approximately 79 months)
Phase 1b and Phase 2: Number of Participants With Markedly Abnormal Laboratory Evaluations | Baseline up to End of Treatment (Up to approximately 79 months)
Phase 1b and Phase 2: Number of Participants With Markedly Abnormal Vital Signs | Baseline up to End of Treatment (Up to approximately 79 months)
Phase 1b and Phase 2: Number of Participants With Clinically Abnormal 12-lead Electrocardiogram (ECG) | Baseline up to End of Treatment (Up to approximately 79 months)
Phase 1b and Phase 2: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | Baseline up to End of Treatment (Up to approximately 79 months)
Phase 1b and 2: Number of Participants With Clinically Significant Abnormal Physical Examination Findings | Baseline up to End of Treatment (Up to approximately 79 months)
Phase 1b and Phase 2, Cmax: Maximum Observed Plasma Concentration of E7389-LF | Phase 1b, Cycle 1 Day 1: 0 to 24 hours, Cycle 1 Days 4 and 8; Phase 2, Cycle 1 Days 1 and 8 (Cycle length = up to 28 days)
Phase 1b and Phase 2: Serum Concentration of Nivolumab | Up to Cycle 13 (each Cycle length = up to 28 days)
Phase 1b and Phase 2, Tmax: Time to Maximum Observed Plasma Concentration (Cmax) of E7389-LF | Phase 1b, Cycle 1 Day 1: 0 to 24 hours, Cycle 1 Days 4 and 8; Phase 2, Cycle 1 Days 1 and 8 (Cycle length = up to 28 days)
Phase 1b and Phase 2, AUC: Area Under the Plasma Concentration-time Curve Over Time From 0 to Last Measurable Concentration of E7389-LF | Phase 1b, Cycle 1 Day 1: 0 to 24 hours, Cycle 1 Days 4 and 8; Phase 2, Cycle 1 Days 1 and 8 (Cycle length = up to 28 days)
Phase 1b and Phase 2, T1/2: Terminal Phase Elimination Half-life of E7389-LF | Phase 1b, Cycle 1 Day 1: 0 to 24 hours, Cycle 1 Days 4 and 8; Phase 2, Cycle 1 Days 1 and 8 (Cycle length = up to 28 days)
Phase 1b and Phase 2, CL: Total Body Clearance of E7389-LF | Phase 1b, Cycle 1 Day 1: 0 to 24 hours, Cycle 1 Days 4 and 8; Phase 2, Cycle 1 Days 1 and 8 (Cycle length = up to 28 days)
Phase 1b and Phase 2, Vd: Volume of Distribution of E7389-LF | Phase 1b, Cycle 1 Day 1: 0 to 24 hours, Cycle 1 Days 4 and 8; Phase 2, Cycle 1 Days 1 and 8 (Cycle length = up to 28 days)
Phase 2: Progression-Free Survival (PFS) | From the first does of the study drug up to the first documentation of disease progression or death due to any cause, whichever comes first (up to approximately 79 months)
  PFS is defined as the time from the date of the first administration of drug to the date of the first documentation of disease progression or death due to any cause, whichever comes first. The PFS will be assessed by investigator based on RECIST version 1.1.

CONTACTS AND LOCATIONS:
Locations (19):
- Japan (19):
  - Eisai Trial Site #13, Nagoya, Aichi-ken
  - Eisai Trial Site #18, Kashiwa, Chiba
  - Eisai Trial Site #2, Kashiwa, Chiba
  - Eisai Trial Site #14, Matsuya, Ehime
  - Eisai Trial Site #4, Kurume, Fukuoka
  - Eisai Trial Site #11, Akashi, Hyōgo
  - Eisai Trial Site #15, Yokohama, Kanaga
  - Eisai Trial Site #3, Sendai, Miyagi
  - Eisai Trial Site #6, Chuo Ku, Osaka
  - Eisai Trial Site #8, Chuo Ku, Osaka
  - Eisai Trial Site #5, Osakasa, Osaka
  - Eisai Trial Site #7, Sakai C, Osaka
  - Eisai Trial Site #17, Suita, Osaka
  - Eisai Trial Site #19, Kitaadachi-gun, Saitama
  - Eisai Trail Site #16, Sunto-g, Shizuo
  - Eisai Trial Site #1, Chuo Ku, Tokyo
  - Eisai Trial Site #10, Koto-Ku, Tokyo
  - Eisai Trial Site #9, Wakayama, Wakaya
  - Eisai Trial Site #12, Kōtoku

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Oshima T, Yamamoto S, Kawakami H, Makino T, Kawazoe A, Masuishi T, Tsushima T, Hirao M, Tsuda M, Hino K, Yamamoto N, Hara H, Kaname S, Matsuoka D, Otake Y, Yasuda K, Takase T, Takashima S, Semba T, Ooki A. Phase 1b/2 study of the liposomal formulation of eribulin (E7389-LF) in combination with nivolumab: Results from the phase 2 esophageal cancer cohort. BJC Rep. 2024 Sep 4;2(1):66. doi: 10.1038/s44276-024-00066-6. PMID 39516370
- [Derived] Kawazoe A, Yamamoto N, Sugimoto N, Kawakami H, Oshima T, Yamaguchi K, Hino K, Hirao M, Kurokawa Y, Kawakami T, Tsuda M, Hara H, Kaname S, Matsuoka D, Otake Y, Yasuda K, Takase T, Takashima S, Semba T, Muro K. Phase II Study of the Liposomal Formulation of Eribulin (E7389-LF) in Combination with Nivolumab: Results from the Gastric Cancer Cohort. Clin Cancer Res. 2024 Apr 1;30(7):1264-1272. doi: 10.1158/1078-0432.CCR-23-1768. PMID 38295160